CLINICAL TRIAL: NCT04384419
Title: Real or Concieved Death Number Perception in Depression, Anxiety and in Schizotypal Personality Disorder Following Covid-19 Pandemic Lockdown
Brief Title: Death Number Perception in Depression, Anxiety, and Schizoypal Personnality in General Population (Covid-19 Pandemic)
Acronym: DeathPercep
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Collaborators: University of Montpellier 3 (Pr. Stéphane Raffard, PhD) (Unknown); University of Reims Champagne-Ardenne (Ali Oker PhD) (Unknown)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0276
Record Dates: First submitted 2020-05-05; First posted 2020-05-12 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Mental Disorder; General Population
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
France has been put on a lockdown for 8 weeks to prevent the spread of the COVID-19 virus between 17/03/2020 and 11/05/2020. During this lockdown, which is likely to have psychopathological repercussions on the population, the public authorities and the media informed the population about the number of deaths occurring each day. While the functioning of autobiographical memory following traumatic events remains a debate in the literature, the impact of the daily announcement of mass deaths on the memory system in the general population and the relationship between long-term memory and delusional thinking in certain psychopathologies have yet to be explored in the literature.

The investigators wish to demonstrate that self-reported recall of recorded deaths may represent this distortion of perception, symptomatic of these pathologies by an on-line questionnaire.

DETAILED DESCRIPTION:
Indeed, it has been reported that under continued stress, delusions and psychotic experiences can occur in the general population. This phenomenon is found in individuals suffering from depression and anxiety and schizotypal personality disorder.

The investigators wish to demonstrate that self-reported recall of recorded deaths may represent this distortion of perception, symptomatic of these pathologies.

Thus, using an online longitudinal questionnaire, the investigators wish to explore :

* how the memory system is impacted by mass deaths over several trimesters in the general population.
* whether the long-term memory of people suffering from depression and anxiety disorders and people suffering from schizotypal personality disorder contains recollection of a distorted pattern in relation to the actual number of deaths.

Primary goals of this project are:

Determine, in the context of mass deaths, the level and proportion of real or conceived recall of the number of deaths in the general population based on cognitive and affective empathy profiles over four trimesters.

Also the investigators want to determine

* the proportion of real or conceived recall numbers of deaths by COVID-19 among people suffering from depression and anxiety in a context of mass death.
* the proportion of real or conceived recall number of deaths by COVID-19 among people with schizotypal personality disorder.
* the dynamics of this real or conceived recall for four trimester following the end of lockdown.

Methodology:

The entire study will be conducted online. Participants will provide their informed consent. At these assessment, they will provide a set of self report measures associated to COVID-19 related psychological aspects especially for depression, anxiety and schizotypal personality.

Subjects can only participate once.

Sample size:

There is no minimum/maximum sample size for this study. The study will remain open for 1 year. The sample size should reach 1000 participants at least.

List of self-report measures:

* Brief Trauma Questionnaire (BTQ)
* COVID-Related Thoughts and Behavioral Symptoms (COV-TaBS)
* Beck Depression Inventory (BDI)
* State and Trait Anxiety Inventory (STAI)
* The Hospital Anxiety and Depression Scale (HAPS)
* Questionnaire of Cognitive and Affective Empathy (QCAE)
* Raine Schizotypal Personality Questionnaire, (SPQ)
* Paranoia Scale

ELIGIBILITY:
Inclusion criteria:

* Individuals from the general population
* French native speacker
* Majority 18 years and more

Exclusion criteria:

* Patient refusing to participate in research

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: General population with self reported depression, anxiety and schizotypal personnality and without mental health conditions
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2020-05-29 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
number of perception distortions | 1 day
  number of perception distortions

SECONDARY OUTCOMES:
Recall number of deaths | 1 day
  Recall number of deaths

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane Raffard, PhD, Principal Investigator — University Hospitals of Montpellier
Locations (1):
- UH Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC